CLINICAL TRIAL: NCT04000048
Title: Phylogenetic Analysis of Intra-tumor Molecular Heterogeneity on a Pilot Series of Diffuse Low-grade Multilobar Gliomas: Tumor Ontogenesis and Therapeutic Implications
Brief Title: Molecular Heterogeneity in Multilobar Low-grade Gliomas
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL18_0376
Record Dates: First submitted 2019-06-25; First posted 2019-06-27 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-06

CONDITIONS: Low-grade Diffuse Glioma
Keywords: Low-grade diffuse glioma; DNA extraction; sequencing

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Biospecimen Retention: Samples With DNA — In this pilot study we chose the fronto-temporal-insular GDBG model to study the intra-tumoral heterogeneity of the low-grade gliomas by exhaustive high throughput sequencing of each of the 3 infiltrated lobes, followed by comparative phylogenetic analysis of the genetic profiles obtained in the 3 locations
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Genetic: sequencing of the complete exome — Once the pathological diagnosis is confirmed (WHO 2016), a tumor fragment will be selected and frozen for each lobe. DNA extraction will be performed for each fragment. The samples (4 different DNAs per GDBG corresponding to the DNA extracted from each of the 3 lobes and the blood DNA) will be sent to the Montpellier Genomix platform for sequencing of the complete exome.

SUMMARY:
Low-grade diffuse glioma (GDBG) are rare tumors of young adults, whose ontogenesis is poorly understood. Patient management is based on the molecular profile defined by two molecular markers : mutations of the IDH genes and chromosomal 1p19q co-deletion. To date, the IDH and 1p19q statuses are determined on a single fragment collected from the tumor. In the case of GDBGs infiltrating several brain lobes, the sampling is done randomly on only one of the infiltrated lobes. An intra-tumoral heterogeneity of genetic alterations has been suggested and would impact management.

Phylogenetic analysis of genetic alterations found, by high throughput sequencing, in each lobe invaded by the same GDBG will make it possible to assess intra-tumoral heterogeneity and to discuss, at a fundamental level, the hypothesis of a single tumor site with secondary diffusion or that of the convergent progression of two or three distinct tumor sites. Clinically, understanding the ontogenesis of GDBGs will improve their management because of the known link between brain location, dominant molecular profile, and prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Be over 18 years old.
* Subject not opposed to participating in the study
* Be scheduled in the operating room for the first surgery of a low-grade diffuse glioma presupposition on the basis of clinical and imaging criteria.
* Confirmation, after histopathological analysis of the resected tumor fragments, of the diagnosis of grade II glioma according to the 2016 WHO classification of brain tumors.

Exclusion Criteria:

* Patient minor, or major under legal protection, or unable to give consent.
* Refusal to participate in the study.
* Pathology diagnosis of grade III glioma according to WHO 2016 classification
* Have received oncology treatment (chemotherapy and or chemotherapy) before the first surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: resected tumor fragments, of the diagnosis of grade II glioma according to the 2016 WHO classification of brain tumors.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Estimated)
Dates: Start 2019-06-24 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Genetic profile | 12 month
  exhaustive high throughput sequencing of each of the 3 infiltrated lobes, followed by comparative phylogenetic analysis of the genetic profiles obtained in the 3 locations

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Gui de Chauliac, Montpellier, France

IPD SHARING:
Plan to Share IPD: No